CLINICAL TRIAL: NCT00374101
Title: Proton Pump Inhibitors in Conjunction to Endoscopic Therapy for Bleeding Peptic Ulcers: a Randomized Clinical Trial of High vs Standard Doses
Brief Title: High Versus Standard Dose of Proton Pump Inhibitors (PPIs) in Peptic Ulcer Bleeding
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Casa Sollievo della Sofferenza IRCCS (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18/2004
Record Dates: First submitted 2006-09-07; First posted 2006-09-08 (Estimated); Last update posted 2007-04-05 (Estimated); Status verified 2007-04

CONDITIONS: Peptic Ulcers; Upper Gastrointestinal Bleeding
Keywords: PPIs,; endoscopic therapy,; peptic ulcers,; upper gastrointestinal bleeding,; non-variceal upper gastrointestinal bleeding
MeSH Terms: conditions — Peptic Ulcer; Gastrointestinal Hemorrhage | interventions — Omeprazole; Pantoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: omeprazole
Drug: pantoprazole

SUMMARY:
High intravenous dosage of Proton Pump Inhibitors is not better than standard dosage in bleeding peptic ulcers successfully treated by endoscopic therapy

DETAILED DESCRIPTION:
The recent Canadian consensus conference on the management of patients with non-variceal upper gastrointestinal bleeding recommends a high regimen of PPIs, consisting in a dosage of 80-mg bolus followed by the 8 mg/H infusion, as being superior to the standard dosage (40 mg twice daily by bolus injection) in conjunction with some type of endoscopic therapy. However, by pooling data fromm studies comparing high doses of PPIs as continuous infusion versus regular doses as intermittent bolus, rebleeding, surgery, and mortality were not significantly different. As the previous conclusion became apparent in a meta-analytical evaluation of only 2 randomized clinical trials, more studies are needed on this topic.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients admitted for upper gastrointestinal bleeding secondary to peptic ulcers that have been successfully treated with endoscopic therapy

Exclusion Criteria:

* Variceal esophageal bleeding
* Concurrent PPI use
* Moribund patients

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450
Dates: Start 2005-01; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Rebleeding rates and surgical needs

CONTACTS AND LOCATIONS:
Overall Officials: Andriulli Angelo, MD, Principal Investigator — Division of Gastroenterology, "Casa Sollievo della Sofferenza", San Giovanni Rotondo, ITALY
Locations (10):
- Italy (10):
  - Division of Internal Medicine, Polla, Salerno
  - Division of Gastroenterology, Caserta
  - DIvision of Gastroenterology, Como
  - Division of Gastroenterology, Cosenza
  - DIvision of Internal Medicine, Ivrea
  - Division of Gastroenterology, Piacenza
  - Division of Gastroenterology, San Giovanni Rotondo
  - Division of Gastroenterology, Torino
  - Division of Gastroenterology, Treviso
  - Division of Gastroenterology, Vasto

REFERENCES:
- [Background] Andriulli A, Annese V, Caruso N, Pilotto A, Accadia L, Niro AG, Quitadamo M, Merla A, Fiorella S, Leandro G. Proton-pump inhibitors and outcome of endoscopic hemostasis in bleeding peptic ulcers: a series of meta-analyses. Am J Gastroenterol. 2005 Jan;100(1):207-19. doi: 10.1111/j.1572-0241.2005.40636.x. PMID 15654802
- [Derived] Andriulli A, Loperfido S, Focareta R, Leo P, Fornari F, Garripoli A, Tonti P, Peyre S, Spadaccini A, Marmo R, Merla A, Caroli A, Forte GB, Belmonte A, Aragona G, Imperiali G, Forte F, Monica F, Caruso N, Perri F. High- versus low-dose proton pump inhibitors after endoscopic hemostasis in patients with peptic ulcer bleeding: a multicentre, randomized study. Am J Gastroenterol. 2008 Dec;103(12):3011-8. doi: 10.1111/j.1572-0241.2008.02149.x. PMID 19086953